CLINICAL TRIAL: NCT06561347
Title: A Phase 2 Multicenter Study of the Combination Zanubrutinib, Bendamustine, and Rituximab in Previously Untreated Waldenström Macroglobulinemia (ZEBRA Trial)
Brief Title: Zanubrutinib, Bendamustine, Rituximab Prev. Untreated WM
Acronym: ZEBRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, Andrew R. Branagan, M.D., Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-294
Record Dates: First submitted 2024-08-05; First posted 2024-08-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: MW; Untreated
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib + Bendamustine + Rituximab (Experimental): Zanubrutinib will be taken orally once daily on days 1-28 of cycles 1-15.
  Bendamustine will be given by intravenous infusion over about 10 to 60 minutes on days 1 and 2 of cycles 1 to 4.
  Rituximab will be given by intravenous infusion over about 30 minutes on day 1 of cycles 1 to 4.
  Drug diaries will be provided to participants to document information about the study treatment being taken.
  Interventions: Drug: Zanubrutinib; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Zanubrutinib — A potent, specific, and irreversible Bruton tyrosine kinase (BTK) inhibitor
  Other Names: BGB-3111
Drug: Bendamustine — Alkylating agent
Drug: Rituximab — Monoclonal antibody

SUMMARY:
The purpose of this study is to determine the very good partial response (VGPR) or better rate in participants with Waldenström macroglobulinemia (WM).

The names of the study drugs involved in this study are as follows: zanubrutinib, bendamustine, and rituximab.

DETAILED DESCRIPTION:
This is multi-center phase 2 of zanubrutinib, bendamustine, and rituximab (ZBR) in previously untreated Waldenström macroglobulinemia (WM).

A phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved bendamustine and rituximab for your specific disease, but it has been approved for other uses.

The U.S. FDA has approved zanubrutinib as a treatment option for your disease.

The combination of zanubrutinib, bendamustine, and rituximab is not approved regimen for Waldenström macroglobulinemia (WM) and is investigational in this study.

Participation is expected for a maximum of 15 cycles and follow-up for up to 5 years.

It is expected that about 50 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of waldenström macroglobulinemia (WM) per the second international workshop on waldenström macroglobulinemia (IWWM2) criteria
* Presence of any MYD88 and CXCR4 mutation status, including MYD88 L265P mutation plus CXCR4 wild type, MYD88 L265P mutation plus CXCR4 mutation, or MYD88 wild type
* Meeting criteria for treatment per IWWM2 criteria. At least one of the following:

  * Constitutional Symptoms (at least one of the following)

    * Recurrent fever
    * Night sweats
    * Fatigue
    * Weight loss
  * Progressive or symptomatic lymphadenopathy or splenomegaly
  * Hemoglobin ≤ 10 g/dL
  * Platelet count ≤ 100 k/uL
  * Hyperviscosity syndrome
  * Symptomatic peripheral neuropathy
  * Systemic amyloidosis
  * Renal insufficiency
  * Symptomatic cryoglobulinemia or cold agglutinemia
* Treatment naive; must have not received any prior systemic therapy for WM
* Participants with suspected or symptomatic hyperviscosity (e.g. nosebleeds, headaches, blurred vision) must undergo plasmapheresis prior to treatment initiation.
* Adults age ≥18
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Women of childbearing potential: Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or practice complete abstinence1 from heterosexual intercourse during treatment and for at least 1 week after the last dose of zanubrutinib or at least 12 months after the last dose of rituximab, whichever is later. FCBP must be referred to a qualified provider of contraceptive methods if needed. Also, FCBP must have a pregnancy check with a negative serum pregnancy test obtained 28 days prior to and confirmed by C1D1.
* Men must agree to use a condom during sexual contact with a female of childbearing potential (FCBP) even if they have had a successful vasectomy 1) while participating in the study; and 2) for at least 1 week following the last dose of zanubrutinib.
* Participants must meet the following organ and marrow function as defined below:

  * Absolute neutrophil count ≥500/mcL believed to be caused by WM bone marrow involvement. Growth factors are not permitted <14 days prior to C1D1.
  * Platelets ≥30,000/mcL believed to be caused by WM bone marrow involvement. Platelet transfusions are not permitted <14 days prior to C1D1.
  * Hemoglobin ≥ 7 g/dL. RBC transfusions are not permitted <14 days prior to C1D1.
  * Total bilirubin ≤ 1.5 X institutional ULN, or ≤3 x institutional ULN with documented liver metastases and/or Gilbert's Disease
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal, or ≤5 X institutional ULN with documented liver metastases
  * Creatinine clearance ≥30 mL/min using the Cockcroft-Gault formula
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, uncontrolled intercurrent illness, or psychiatric illness/social condition that would prevent the participant from signing the informed consent form
* Female participants who are pregnant, breastfeeding, or planning to become pregnant or breastfeed while enrolled in this study
* Participants with known CNS involvement by WM
* Participants with known history of Human Immunodeficiency Virus (HIV)
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below:

  * Hepatitis B virus (HBV): Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (antiHBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation before enrollment. Patients who are hepatitis B PCR positive will be excluded.
  * Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before enrollment. Patients who are hepatitis C RNA positive will be excluded.
* Concurrent systemic immunosuppressant therapy. Systemic steroids at doses <20mg prednisone per day are permitted.
* Active and/or ongoing autoimmune anemia and/or autoimmune thrombocytopenia (eg, idiopathic thrombocytopenia purpura).
* Concurrent administration of warfarin or warfarin derivatives.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Active uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the Investigator and the Sponsor makes it undesirable for the patient to participate in the trial. Screening for chronic conditions is not required. Active uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the Investigator and the Sponsor makes it undesirable for the patient to participate in the trial. Screening for chronic conditions is not required.
* Major surgery within 4 weeks of first dose of study drug.
* History of severe bleeding disorder such as hemophilia A, hemophilia B, or history of spontaneous bleeding requiring blood transfusion or other medical intervention. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.
* Participants with inability to swallow pills.
* Inability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of the study participation.
* Any uncontrolled or significant cardiovascular disease defined as:

  * Unstable angina within 3 months before screening, or
  * History of myocardial infarction within 6 months prior to planned start of zanubrutinib, or
  * Previously documented left ventricular ejection fraction (LVEF) by any method of ≤ 45% in the 12 months prior to planned start of zanubrutinib; assessment of LVEF via echocardiogram or multigated acquisition (MUGA) scan during Screening should be performed in selected patients as medically indicated, or
  * Any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or
  * Uncontrolled or symptomatic arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes)
* Participants with a known hypersensitivity to any of the excipients of Zanubrutinib, Rituximab, or Bendamustine.
* Participants with a history of non-compliance to medical regimens, which will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs.
* Prior malignancy within the past 3 years, except for curatively treated basal or squamous cell skin cancer, non-muscle-invasive bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 prostate cancers.
* Severe or debilitating pulmonary disease.
* Ongoing alcohol or drug addiction or any psychiatric condition(s) which would compromise ability to comply with study procedures.
* Ongoing use of a strong CYP3A inducer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Very Good Partial Response (VGPR) or Better Response Rate | Day 1 to 5 years post treatment
  Assessed using 11th International Workshop on Waldenstrom's Macroglobulinemia (IWWM11) criteria. All participants will be gauged for very good partial response (VGPR) rate or better.

SECONDARY OUTCOMES:
Treatment Related Adverse Events | Day 1 to 5 years post treatment
  Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All participants will be followed and assessed for safety and tolerability of the protocol therapy.
Overall Response Rate | Day 1 to 5 years post treatment
  Assessed per 11th International Workshop on Waldenstrom's Macroglobulinemia (IWWM11) criteria. All participants by mutational status will be monitored for minor response (MR), partial response (PR), very good partial response (VGPR), and complete response (CR).
Major Response Rate | Day 1 to 5 years post treatment
  Assessed per 11th International Workshop on Waldenstrom's Macroglobulinemia (IWWM11) criteria. All participants by mutational status will be monitored for partial response (PR), very good partial response (VGPR), and complete response (CR).
Complete Response Rate | Day 1 to 5 years post treatment
  Assessed per 11th International Workshop on Waldenstrom's Macroglobulinemia (IWWM11) criteria. All participants by mutational status will be monitored for having resolution of Waldenstrom's Macroglobulinemia (WM) related symptoms, normalization of serum Immunoglobulin M (IgM) levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly. A complete response requires reconfirmation demonstrating normal serum IgM levels, and absence of IgM paraprotein by immunofixation by a measurement repeated at least 2 weeks later.
Median Time to Response | Day 1 to 5 years post treatment
  All participants by mutational status will be assessed per 11th International Workshop on Waldenstrom's Macroglobulinemia (IWWM11) criteria.
Median Time to Major Response | From Day 1 until date of major response is first documented, assessed up to 5 years post treatment
  All participants by mutational status will be assessed per 11th International Workshop on Waldenstrom's Macroglobulinemia (IWWM11) criteria.
Median time to Next Treatment | From Day 1 until date of next line of therapy is first documented, assessed up to 5 years post treatment
  The duration of time from the initiation of study treatment to the date of commencement of the next line of therapy.
Progression-Free Survival | From Day 1 until date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 5 years post treatment
  The duration of time from start of treatment to time of objective disease progression or death. Median, 2-year and 4-year landmark progression free survival (PFS) analysis will be determined.
Overall Survival | From Day 1 until date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 5 years post treatment
  The duration of time from start of treatment to time of death or last follow-up. Median, 2-year and 4-year landmark overall survival (OS) analysis will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Branagan, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Colorado Blood Cancer Institute (CBCI), Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation